CLINICAL TRIAL: NCT01015183
Title: Prevention High Dose Chemotherapy Induced Mucositis by Using Zinc Sulfate
Brief Title: Prevention Chemotherapy Induced Mucositis by Zinc Sulfate
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Mahdi Jalili MD / Hematology-Oncology and SCT Research Center, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HORCSCT-0904
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Mucositis; Bone Marrow Transplantation
Keywords: Mucositis; Bone Marrow Transplantation; BMT; HSCT
MeSH Terms: conditions — Mucositis | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Received Zinc Sulfate
  Interventions: Drug: Zinc Sulfate
- Control (Placebo Comparator): Control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc Sulfate — Zinc Sulfate: 100 mg of zinc element, per day, bid for two weeks start with chemotherapy
  Arms: Intervention
Drug: Placebo — Placebo: as the same of intervention group
  Arms: Control

SUMMARY:
In this double blinded randomized study we evaluate effect of Zinc sulfate for prevention mucositis due to high dose chemotherapy in the patients undergoing bone marrow transplantation whose received Busulfan and/or Cyclophosphamide. Patients randomized in two groups: intervention and control with balanced block randomization method. Intervention group received Zinc sulfate immediately after start conditioning regimen and continued for two weeks. Control group received placebo at the same manner. Prevalence and severity of mucositis will be compared in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing bone marrow transplantation
* Signed informed consent

Exclusion Criteria:

* Unable take drug (or placebo) orally

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The effect of Zinc Sulfate on prevention of mucositis in patients undergoing bone marrow transplantation | 1 year

SECONDARY OUTCOMES:
Evaluation of Zinc Sulfate concentration | 1 year
Evaluation of Zinc Sulfate advance effects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Molouk Hadjibabaie, PhD, Principal Investigator — Hematology-Oncology and SCT Research Center
Locations (1):
- Hematology-Oncology & SCT Research Center, Tehran, Tehran Province, Iran